CLINICAL TRIAL: NCT01827501
Title: Can Perioperative Goal Directed Hemodynamic Management Reduce the Incidence of Delirium in Older Patients After Major Non-cardiac Surgery?
Brief Title: Avoidance of Delirium in Older Patients After Major Non-cardiac Surgery
Acronym: ADOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADOM
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Delirium
Keywords: postoperative delirium; hemodynamic management; goal directed therapy
MeSH Terms: conditions — Delirium; Emergence Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group GDT (Experimental): Goal-directed Management according to pulse contour analysis (PulsioflexTM Monitoring)
  Interventions: Device: PulsioflexTM Monitoring
- Group Co (No Intervention): Conventional fluid management

INTERVENTIONS:
Device: PulsioflexTM Monitoring — Fluid and catecholamine management according to PulsioflexTM measurements
  Arms: Group GDT

SUMMARY:
This study is designed to compare the incidence of postoperative delirium in older patients after major non-cardiac surgery with different perioperative hemodynamic managements: a goal directed hemodynamic management group and a control group

DETAILED DESCRIPTION:
Delirium is a common postoperative complication in the elderly. The incidence depends on several factors like the comorbidities of the patient and the type of surgery. Mortality is almost twofold increased after two years for patients suffering from delirium after surgery. Different studies showed that with a multimodal strategy it was possible to reduce the risk of delirium. As several different organ systems are involved in the development of delirium the patient's hemodynamic state seems to be important and is a target point of intervention. Also sufficient perfusion and oxygen delivery is essential in order to avoid impairment of the brain. Recent studies showed that goal directed hemodynamic management can reduce all kind of postoperative complications and improve outcome. However, whether the use of goal-directed hemodynamic management also improves the neurological outcome and reduces the rates of postoperative delirium has not been studied yet.

Aim of this study is to investigate the impact of goal directed hemodynamic management using pulse contour analysis on the incidence of delirium in older patients undergoing non-cardiac surgery, presenting with an intermediate to high risk for delirium. This risk will be assessed preoperatively using a score suggested by Marcantonio.

Patients will be randomized in one of two groups, the goal-directed therapy group and the control group. In the goal-directed therapy (GDT) group hemodynamic management is performed according to an established algorithm obtained by pulse contour analysis. To prove our theory that goal-directed therapy influences the brain by increasing oxygen supply we will use near infrared spectroscopy, which is safe and non-invasive, in our patients. The hemodynamic management is continued in the recovery room or at the intensive care unit according to the mentioned algorithm. The intervention will be terminated as soon as patients fulfil the standard criteria for discharge from recovery room or intensive care.

In the control group hemodynamic management is performed according to heart rate and blood pressure without using extended monitoring.

As the actual incidence has a significant impact on the number needed per group, we are going to perform an interims analysis after 100 included patients according to the O'Brian-Fleming technique. Is the difference of delirium between the two groups significant with an α < 0,002 the study will be finished. Otherwise, the sample size needed per group will be determined assuming an α = 0,048, a two-tailed test and a power of 80%.

UPDATE 19-10-2016:

The interims-analysis of incidences after 100 patients revealed, that 86 patients per group will be needed (α = 0,048, power 80%).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Risk of perioperative delirium (Marcantonio) ≥6

Exclusion Criteria:

* Emergency surgery
* Valvular disorders grad II or higher
* History of major aortic surgery
* Major aortic surgery
* Repeated surgery (within 30 days before)
* Neurosurgery

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 172 (Actual)
Dates: Start 2013-04; Primary Completion 2019-12 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium until day 7 (CAM-Score and clinical diagnosis) | Before induction of anesthesia until 7 days after surgery
  Delirium according to CAM-Score and clinical diagnosis

SECONDARY OUTCOMES:
Factors defining delirium | 7 days
  Duration of delirium, total amount of haloperidol administered
Short-term cognitive impairment | 7 days
  Mini Mental State on day 7
Mortality | 1 year
  in-hospital mortality, mortality after one year
Influence on brain oxygen saturation | until discharge from recovery room/ICU
  Influence of GDT on the frontal oxygen saturation of the brain assessed with Near-InfraRed-Spectroscopy (NIRS)-Monitoring
Intra- and postoperative Measurements | Until discharge
  Time until discharge, total fluids and amount of catecholamines administered, incidence of overall postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Jungwirth, MD, Principal Investigator — Klinik für Anaesthesiologie Technische Universität München
Locations (1):
- Klinik für Anästhesiologie Klinikum Rechts der Isar, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marcantonio ER. Postoperative delirium: a 76-year-old woman with delirium following surgery. JAMA. 2012 Jul 4;308(1):73-81. doi: 10.1001/jama.2012.6857. PMID 22669559
- [Derived] Fuest KE, Servatius A, Ulm B, Schaller SJ, Jungwirth B, Blobner M, Schmid S. Perioperative Hemodynamic Optimization in Patients at Risk for Delirium - A Randomized-Controlled Trial. Front Med (Lausanne). 2022 Jul 13;9:893459. doi: 10.3389/fmed.2022.893459. eCollection 2022. PMID 35935775